CLINICAL TRIAL: NCT02172937
Title: Decidual Stromal Cells as Treatment for Acute Graft Versus Host Disease
Brief Title: Decidual Stromal Cells as Treatment for Acute Graft Versus Host Disease, a Phase 1-2 Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Olle Ringdén, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSCGVHD002
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Graft vs Host Disease
Keywords: Stem Cell Transplantation; Decidual Stromal Cells
MeSH Terms: conditions — Graft vs Host Disease | interventions — Serum Albumin, Human

ARMS (2):
- Decidual Stromal Cells as last line treatment (Experimental): Patients with therapy-refractory GVHD and on calcineurin inhibitor and high dose corticosteroids without any signs of improvement will be given DSCs to evaluate a possible effect. DSCs will be thawed from the freezer in plasma.
  Interventions: Biological: Decidual Stromal Cells thawed in plasma
- Decidual Stromal Cells (Active Comparator): Patients with therapy-refractory GVHD and on calcineurin inhibitor and high dose corticosteroids will be given DSCs as early as possible at one or more occasions at weekly intervals dependent on clinical response. DSCs will be thawed from the freezer in plasma.
  Interventions: Biological: Decidual Stromal Cells thawed in human albumin

INTERVENTIONS:
Biological: Decidual Stromal Cells thawed in plasma
  Arms: Decidual Stromal Cells as last line treatment
Biological: Decidual Stromal Cells thawed in human albumin
  Arms: Decidual Stromal Cells

SUMMARY:
The purpose of this study is to evaluate safety and efficacy using decidual stromal cell therapy for graft versus host disease after allogeneic hematopoietic stem cell transplantation. The hypothesis to be tested is that the cells are safe to infuse and that they have a positive clinical effect.

DETAILED DESCRIPTION:
Patients with GVHD grade 2-4, will receive decidual stromal cells at approximately 1-2x10^6 cells/kg at one or more occasions dependent on clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Acute graft versus host disease grade 2-4.
* Are on calcineurin inhibitor and high dose corticosteroids.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Actuarial survival at six months after first DSC infusion | 6 months after inclusion

SECONDARY OUTCOMES:
Response at 28 days after onset of graft versus host disease | 28 days after inclusion
  Response will be measured as:
  * Partial response (PR) if the patient has improved one grade in the overall GvH.
  * Complete response (CR) if the patient is free of GvH.
  * Non responder (NR) if the patient does not improve after treatment.
Response at 84 days after onset of graft versus host disease | Up to 84 days after inclusion
  Response will be measured as:
  * Partial response (PR) if the patient has improved one grade in the overall GvH.
  * Complete response (CR) if the patient is free of GvH.
  * Non responder (NR) if the patient does not improve after treatment.
Response at 168 days after onset of graft versus host disease | Up to 168 days after inclusion
  Response will be measured as:
  * Partial response (PR) if the patient has improved one grade in the overall GvH.
  * Complete response (CR) if the patient is free of GvH.
  * Non responder (NR) if the patient does not improve after treatment.
Side effects | Up to 6 months after inclusion
  Adverse effects related to the treatment.
Incidence of severe infections | Up to one year after inclusion
  Severe bacterial, viral and fungal infections.
Disease free survival | Up to one year after inclusion
  Survival free from relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Olle Ringdén, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Erkers T, Nava S, Yosef J, Ringden O, Kaipe H. Decidual stromal cells promote regulatory T cells and suppress alloreactivity in a cell contact-dependent manner. Stem Cells Dev. 2013 Oct 1;22(19):2596-605. doi: 10.1089/scd.2013.0079. Epub 2013 Jul 2. PMID 23701127
- [Result] Ringden O, Erkers T, Nava S, Uzunel M, Iwarsson E, Conrad R, Westgren M, Mattsson J, Kaipe H. Fetal membrane cells for treatment of steroid-refractory acute graft-versus-host disease. Stem Cells. 2013 Mar;31(3):592-601. doi: 10.1002/stem.1314. PMID 23307526
- [Derived] Sadeghi B, Remberger M, Gustafsson B, Winiarski J, Moretti G, Khoein B, Klingspor L, Westgren M, Mattsson J, Ringden O. Long-Term Follow-Up of a Pilot Study Using Placenta-Derived Decidua Stromal Cells for Severe Acute Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2019 Oct;25(10):1965-1969. doi: 10.1016/j.bbmt.2019.05.034. Epub 2019 Jun 4. PMID 31173898